CLINICAL TRIAL: NCT01643694
Title: Randomized Controlled Trial Evaluating the Effect of An Individualized Electronic Intervention to Promote Resilience, Meaning, and Engagement for Physicians
Brief Title: Individualized Electronic Intervention to Promote Work Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Liselotte (Lotte) N. Dyrbye, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 12-004566
Record Dates: First submitted 2012-06-27; First posted 2012-07-18 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Resilience; Meaning in Work; Engagement at Work

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic intervention (Experimental): Completion of 1 self-directed activity from an electronically provided list sent to them weekly for 10 consecutive weeks
  Interventions: Behavioral: Electronic intervention suggesting behavioral activity
- control group (No Intervention): Completion of baseline and 3 mo survey

INTERVENTIONS:
Behavioral: Electronic intervention suggesting behavioral activity — 3.6 Those randomized to the intervention will be asked to choose 1 self-directed activity from an electronically provided list sent to them weekly for 10 consecutive weeks. Each activity will take less than 5 minutes to complete. They will also answer 3-5 questions weekly (items taken from the survey items list submitted).
  Arms: Electronic intervention

SUMMARY:
To determine if physicians who complete brief tasks intended to promote meaning in work and job satisfaction, foster teamwork and social support at work, nuture personal relationships and work-life balance, recognize and build on personal strengths, encourage effective problem solving, and promote positive emotions have improved resilience, meaning in work, and engagement at work.

ELIGIBILITY:
All physicians at Mayo Clinic

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Job satisfaction | baseline to 3 month
  Physician Job Satisfaction Scale and Empowerment at Work Scale

SECONDARY OUTCOMES:
Well-being | Baseline to 3 months
  Maslach Burnout Inventory, 2-item Primary Care Evaluation of Mental Disorders [PRIME MD]), Medical Outcomes Study Short Form [SF-8]; Linear Analogue Scales Assessment Well-being Survey [LASA]), 10-item Perceived Stress Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte Dyrbye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860